CLINICAL TRIAL: NCT02024126
Title: Exercise Therapy in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Västervik hospital (Västervik, Sweden; recruiting clinical unit) (Unknown); City Rehab (Luleå, Sweden; recruiting clinical unit) (Unknown); Moholt Fysioterapi (Trondheim, Norway; recruiting clinical unit) (Unknown); Rosenborg klinikken (Trondheim, Norway; recruiting clinical unit) (Unknown); Frisk 3 (Mosjöen, Norway; recruiting clinical unit) (Unknown); NTNU (Norwegian Univ Science and Tech), Faculty of Health and Social Sciences (Unknown)
Responsible Party: Principal Investigator, Björn O. Äng, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOM-TOR-2009; KI-TOM-TOR-2013 (Other: 0)
Record Dates: First submitted 2013-12-17; First posted 2013-12-31 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Exercise therapy; RCT; Intervention; Knee pain; Muticenter; Knee function
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dosage exercise therapy (Experimental): The high-dosage exercise treatment will be conducted under supervision of experienced physiotherapists, and it follows an exercise protocol previously described as Medical Exercise Therapy, MET. The regimen contains different semi-global and local exercises for the knee. To be able to reach a high number of repetitions despite ongoing pain, the principle of de-loading (reducing weight) will be applied. The use of de-loading allows high number of repetitions nearly or entirely pain free. Later, as the patient improves and tolerates increased loading, the exercises are adapted to be more functional, using closed chain exercises without de-loading the body. Each of the exercises will be performed in 3 sets of 30 repetitions with 30-60s rest in between. Global exercises using a stationary bike will be performed three times during one treatment-session; first 20 minutes as global pain modulation, ten minutes in the middle of the treatment, and then ten minutes at the end of the treatment.
  Interventions: Other: Exercise therapy
- Lower dosage exercise therapy (Active Comparator): Patients in the comparison-/control group will perform six exercises, of which, five will be in 2 sets of 10 repetitions combining local and semi-global exercises, again using the principle of de-loading. The five semi-global and local exercises are the same as performed in the MET-group, and the regimen will be supervised in the same manner as for the MET-group. The therapy starts with 10 minutes using a stationary bike, and the same principles will be applied as for the MET-group regarding grading and follow-up with exercises and adjusting the exercises so that they are performed close to pain-free.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — Exercise therapy

SUMMARY:
Osteoarthritis (OA) is one of the most common form of chronic diseases in the adult population, and approximately 800 000 people in Sweden (population of 9 million people) suffer from this disease, which causes joint pain, stiffness, swelling, loss of function and sick leave. There is increasing evidence that exercise therapy is effective for patients with knee OA. However, there is little knowledge on long-term effects and what type of exercises dosage is most effective. In this present clinical trial, which is a Nordic collaborative project with researchers from different research groups in Sweden and Norway, we intend to investigate short and long-term effects comparing high dosage exercise therapy (each treatment lasting 80 to 90 min) vs. a relatively low dosage exercise program (25 to 30 min) in patients diagnosed with knee OA. Patients in both intervention groups receive three treatments a week for 12 weeks making a total of 36 treatments. Primary outcome is pain-ratings and function (The Knee Injury and Osteoarthritis Outcome Score (KOOS)). Secondary outcome concerns various health-ratings and objective functional tests. Regarding predictors for outcome, we plan also to investigate different psychosocial variables as well as patient's beliefs regarding exercise. Feasibility of how high-dose exercise therapy actually works in primary care health care settings is also planned to be reported.

Patients are being assessed by blinded assessor at inclusion, at end of intervention (3 mo), and at six and 12 mo after end of treatment. We plan to include a total of 200 subjects from primary health care settings, two in Norway and two in Sweden, with radiographic-verified knee OA with knee pain and decreased function. The patients have to be within the 45 to 85 age group. Patients are excluded if they have been scheduled for knee surgery or have some other form of illness/disease that limits the exercise tolerance (e.g. heart disease or systemic/metabolic diseases or chronic obstructive airways disease). A major goal is to grade exercises so that they are performed pain-free or close to pain-free in both intervention groups. The principle of deloading is used to meet this goal using a high number of repetitions in sets as pain modulation. The results from this study will give new information about the effectiveness of graded exercise therapy in patients with knee OA, and new knowledge if outcome can be related to the exercise dosage performed.

DETAILED DESCRIPTION:
Osteoarthritis is one of the most common form of chronic diseases in the adult population, and approximately 800 000 people in Sweden (population of approximately 9 million people) suffer from this disease, which causes joint pain, stiffness, swelling, loss of function and sick leave. Studies from Sweden, United Kingdom (UK) and USA show that costs for osteoarthritis are about 1-2.5 % of GDP. With increasing life expectancies and the general decrease in physical activity in western industrialized countries, it is expected that more people will suffer from this disease. In a recent international literature review of clinical studies on the effectiveness of exercise therapy, the authors concluded that there is some evidence that therapeutic exercise is effective reducing knee pain and improving activities of daily living. In a compilation of scientific studies by the Swedish Council on Technology Assessment in Health Care (SBU), it was concluded that strength and flexibility exercises resulted in positive short-term effects compared to information only. However, there is currently no scientific study that has evaluated dose-response effects of exercise therapy. To improve life quality for individuals with osteoarthritis and the use of exercise therapy in primary and secondary health care settings, research on dose response effects in patients with osteoarthritis is important. This view is supported by various systematic reviews including the report from Swedish Council on Health Technology Assessment (SBU) latest compilation.

Exercise dosage is a factor of exercise frequency, intensity and duration. Recent clinical trials show positive effects at both short term-(end of intervention) and at long term follow ups (6- and 12 months), in favor of high repetitive high dosage exercise therapy compared to a relatively lower exercise dosage in patients with long-term subacromial pain and in patients with long term patello femoral pain syndrome. Compared to treatment as usual, exercise therapy has also been shown to be effective as postsurgical rehabilitation after arthroscopic surgery in patients with knee pain with a verified ruptured mensicus. In this present clinical trial, which is a Nordic collaborative project with researchers from different research groups in Sweden and Norway, we intend to investigate short and long-term effects comparing high dosage exercise therapy versus a low repetitive low dosage exercise program in patients diagnosed with knee osteoarthritis. Primary outcome is pain (VAS) and knee function (The Knee Injury and Osteoarthritis Outcome Score (KOOS)). Since it is unknown which patients will respond to the different exercise dosages, we will also look at different prognostic factors related to patient's beliefs regarding exercise therapy as well as different psychosocial variables as anxiety, depression, fear of movement, catastrophizing, life satisfaction and level of self-efficacy. We hope this study will increase our knowledge regarding positive and negative predictors for outcome.

Thus, the main aim of the study is to evaluate two modes of exercise therapy focusing on exercise dosage; 1) exercise therapy with an exercise dosage lasting 80 - 90 minutes duration at each treatment compared to; 2) low dosage exercise therapy (conventional exercise treatment) lasting 20-30 minutes at each treatment) in patients with long-term knee osteoarthritis. All patients in both intervention groups will receive three treatments a week for 12 weeks making a total of 36 treatments. Physiotherapists at four different intervention centers will treat patients from both exercise interventions. Assessments will be performed at inclusion, after end of treatment, and at six and 12 months follow up. Objective tests (20 meter walk test, sit to stand in 30 seconds and maximum number of single knee flexion/extension in 30 seconds) is tested out at inclusion and at end of treatment. The testers are blinded regarding intervention group. Questionnaires are filled out by the patient at inclusion, end of treatment, at six and 12 months follow up. To assess when possible clinical interesting changes start to occur during the three month treatment period, patients are filling out KOOS (function) and VAS (pain) after every 6th treatment making a total of six measurements during the intervention period.

Patients are recruited from primary care health care settings in Västervik and Luleå in Sweden and in Trondheim and Mosjöen in Norway. Patients are informed about the project both verbally and also through written information. Based on this information, patients that would like to participate in the project, contact the local investigation center to be assessed for possible inclusion. We are planning to include a total of 200 patients with radiographic-verified knee osteoarthritis with knee pain and decreased function. The patients have to be within the 45 to 85 age group, come for three treatments a week, a total of 36 treatments for 12 weeks, and must not have had any treatments or organized form of exercise therapy for their knee pain the last three months. Patients are also excluded if they have been scheduled for knee surgery or have some other form of illnesses/disease that limits exercise tolerance (e.g. heart disease or systemic/metabolic diseases or chronic obstructive airways disease). Patients that fulfill the inclusion criteria will be randomized either to high dosage medical exercise therapy or low dosage exercise therapy.

Each treatment in the high dosage group (also called "Medical Exercise Therapy, MET) consist of 20 minutes global exercise (e.g. stationary cycling), then four local knee exercises either open or closed chain performing three sets of 30 repetitions or five minutes continuous repetitions, then another five minutes cycling followed by another four local knee exercises three sets of 30 repetitions or five minutes continuous repetitions and finishing with 10 minutes cycling. Each treatment lasts 80 to 90 minutes. The patients in this group shall also perform one home exercise every day performing three sets of five minutes deloaded knee extension with therabands. In the low dosage exercise group the patients perform a total of five exercises; 10 minutes warm up using a stationary bicycle, then four different knee exercises performing two sets of 10 repetitions. Each treatment last 20 to 30 minutes.

For all patients in both intervention groups the same methods are applied for testing out exercises at the start of the treatment, and for grading exercises during the treatment period. A major goal is to grade exercises so that they are performed pain-free or close to pain-free in both intervention groups. The exercises are standardized for both exercise programs, however individualized and graded continuously in relation to the patient's clinical status. All treatments are carried out under the supervision of experienced and skilled physiotherapists.

The treating physiotherapists are instructed to be neutral regarding their beliefs of which treatment they believe is most effective informing the patient; in this study we are comparing two different forms of exercise therapy and we do not know if one exercise mode is better than the other or if they have equal effects.

The theoretical basis for MET and the exercise progressions have been described in scientific articles and book chapters. Self-assessed pain, function and quality of life are monitored both during treatment and after treatment, and at six and 12 months follow-up. Prognostic markers evaluated by following analyze background information and early test results relate to the long-term treatment outcome. Analysis of cost-effectiveness will be done using the incremental cost-effectiveness ratio (ICER), in order to provide a single measure for weighing costs against effects of the exercise dosage interventions. An assessment will also be made for the cost per quality-adjusted life year (QALYs).

Our project team has extensive experience with the practical implementation of clinical controlled studies and analytical methodology linked to registries and health economic cost estimates. From this study we expect increased knowledge of whether clinical outcomes from exercise therapy may be related to exercise dosage and how exercise therapy need to be individualized according to the patient's history, clinical picture and coping strategies obtaining. In a recent report from the Swedish Council on Health Technology Assessment (SBU) they requested such data evaluating both the effects of exercise treatment analyzes that support personalized rehabilitation.

The results from this study will give new information about the effectiveness of exercise therapy for patients with knee osteoarthritis, and new knowledge if outcome can be related to the dosage of exercise performed.

ELIGIBILITY:
Inclusion Criteria:

* age 45-85 yrs with an x-ray verified knee osteoarthritis with pain and decreased function.

Exclusion Criteria:

* Inflammatory joint disease, current anterior cruciate ligament injury, hip symptoms more aggravating than the knee symptoms, scheduled to have knee replacement surgery within 12 months, and co-morbidities not allowing exercise like cardiovascular, respiratory, systemic, or metabolic conditions limiting exercise tolerance.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2013-12; Primary Completion 2017-08-31 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Self-assessed function (KOOS) at three months follow-up (other follow-ups with this measure includes six and 12 months follow-up). | At three months follow-up, i.e. after end of treatment (primary end point). In addition, during the intervention period, the KOOS are assessed after every sixth treatment meaning after 2, 4, 6, 8, 10 weeks, as well as at 6 and 12 months follow-up.
  The primary outcome measure is the disease specific Knee injury and Osteoarthritis Outcome Score (KOOS). The KOOS assesses the patients' self-report of pain, other symptoms, activities of daily living, sport and recreation function, and knee-related quality of life, answering 42 questions which take about 10 minutes to complete. The KOOS is scored from 0 to 100, separately for each subscale, 0 indicating extreme problems and 100 indicating no problems.

SECONDARY OUTCOMES:
Patient Satisfaction | After treatment at three months follow-up
  Reflects patients satisfaction with treatment, using self-rated Patient Satisfaction scale (6 point scale)
Anxiety and depression | At baseline, at three months, at six months and at one year follow-up
  Hospital Anxiety and Depression scale (HAD), measured with HAD questionnaire.
Catastrophizing | At baseline, at three months, at six months and at one year follow-up
  Patients level of catastrophizing using Catastrophizing Scale (PCS)
Tama Scale of Kinesiophobia (TSK) | At baseline, at three months, at six months and at one year follow-up
  Patients beliefs and attitudes regarding pain and physical activity using the self-rated Tampa Scale of Kinesiophobia (TSK).
Change from baseline in self assessed pain using a visal analogue scale (VAS) at three months follow-up (other follow-ups with this measure includes six and 12 months follow-up) | At three months follow-up, i.e. after end of treatment. In addition, during the intervention period, the VAS are assessed after every sixth treatment meaning after 2, 4, 6, 8, 10 weeks, as well as at 6 and 12 months follow-up.
  Pain is measured using a 100 mm long line with no pain at 0 and the worst imaginable pain at 100 mm. The patient make a line vertically on the 100mm long line according to the pain experience.

OTHER OUTCOMES:
20 min walk test. | At inclusion and at three months follow-up, i.e. after end of treatment
  20 m walk test. Patients are asked to walk between two visible lines marked on the floor; first with their usual pace, and then at the maximal pace the patient feel secure.
30s Maximal Repeated Unilateral Knee Bending test | At inclusion and at three months follow-up, i.e. after end of treatment
  The test evaluates the maximum number of knee bends in 30 seconds performed on one leg in standing. Both (legs)knees are tested
the Five Time Repeated Chair Stands. | At inclusion and at three months follow-up, i.e. after end of treatment
  The patient is seated in a standard chair (seat height, 40 cm) without armrests, and is instructed to rise to a fully erect standing position five times as fast as possible without using their hands. Outcome is time the patient use to perform the five time repeated chair stands.
Pain and sensory threshold assessment. | At inclusion and at three months follow-up, i.e. after end of treatment
  Using a Cefar PainMatcher, a pain and sensory threshold assessment tool, subjects will have their baseline and pos-treatment pain thresholds recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Björn O Äng, Assoc.prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
This is currently not planned, but may be necessary depending on the requirements of future financiers (it will then be necessary to compliment our ethical application). Data monitoring ("yes", as indicated above) concerns an external person that will monitor our data, and log results in a notebook

REFERENCES:
- [Derived] Rugelbak GM, Torstensen TA, Paulsberg F, Grooten WJA, Osteras H. Does exercise adherence influence outcome in knee osteoarthritis? - a secondary analysis of a superiority randomized controlled trial. Physiother Theory Pract. 2025 Oct 31:1-15. doi: 10.1080/09593985.2025.2579576. Online ahead of print. PMID 41170926
- [Derived] Torstensen TA, Osteras H, LoMartire R, Rugelbak GM, Grooten WJA, Ang BO. High- Versus Low-Dose Exercise Therapy for Knee Osteoarthritis : A Randomized Controlled Multicenter Trial. Ann Intern Med. 2023 Feb;176(2):154-165. doi: 10.7326/M22-2348. Epub 2023 Jan 24. PMID 36689746
- [Derived] Torstensen TA, Grooten WJA, Osteras H, Heijne A, Harms-Ringdahl K, Ang BO. How does exercise dose affect patients with long-term osteoarthritis of the knee? A study protocol of a randomised controlled trial in Sweden and Norway: the SWENOR Study. BMJ Open. 2018 May 5;8(5):e018471. doi: 10.1136/bmjopen-2017-018471. PMID 29730615